CLINICAL TRIAL: NCT03563040
Title: A Prospective, Multicenter, Single-Arm Cohort Study of Photopheresis in the Treatment of Erythrodermic MF and SS
Brief Title: Study of Photopheresis in the Treatment of Erythrodermic MF and SS
Acronym: PROMPT
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of feasibility
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Collaborators: Mallinckrodt (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EORTC-1636-CLTF; 2018-001685-42 (EudraCT Number)
Record Dates: First submitted 2018-05-25; First posted 2018-06-20 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2021-08

CONDITIONS: Lymphoma, T-Cell, Cutaneous; Mycosis Fungoides/Sezary Syndrome
MeSH Terms: conditions — Lymphoma, T-Cell, Cutaneous; Mycosis Fungoides; Sezary Syndrome | interventions — Methoxsalen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Methoxsalen with the THERAKOS CELLEX Photopheresis System (Experimental): Treatment will be performed according to a predefined protocol based on the consensus guidelines in patients with MF/SS. Treatment should be administered for one year unless confirmed disease progression or unless other criteria for treatment discontinuation are met as specified in the protocol.
  Interventions: Drug: Methoxsalen; Device: THERAKOS CELLEX Photopheresis System

INTERVENTIONS:
Drug: Methoxsalen — Methoxsalen is used in conjunction with the THERAKOS CELLEX Photopheresis System.
  During each photopheresis treatment with methoxsalen, the dosage of methoxsalen is calculated according to the treatment volume (which is displayed on the display panel of the instrument) using the formula:
  Treatment volume x 0.017 ml of methoxsalen (20 µg/mL) for each treatment For example: Treatment volume = 240 mL x 0.017 = 4.1 mL of methoxsalen (20 µg/mL)
  Other Names: Uvadex
Device: THERAKOS CELLEX Photopheresis System — Methoxsalen is used in conjunction with the THERAKOS CELLEX Photopheresis System.

SUMMARY:
PROMPT: a study of photopheresis for the treatment of erythrodermic mycosis fungoides and Sézary syndrome

For this study, the investigators invite patients suffering from erythrodermic mycosis fungoides (MF) and Sézary syndrome (SS) whose skin symptoms have not responded to other types of treatment prescribed by their doctors (symptoms came back or got worse) as well as patients that never received any treatment.

Patients will be treated with photopheresis every two weeks for the first three months, thereafter once monthly. One treatment cycle consists of 2 day treatment in a row. After 6 months of treatment, treatment can be given every 5 to 8 weeks.

During the photopheresis procedure, the patient's blood is collected into a specialized machine (THERAKOS CELLEX) that separates the white blood cells from the other blood components. The other blood components are returned to the patient and white blood cells are then treated with the drug methoxsalen, which makes them sensitive to ultraviolet light. The treated white blood cells are exposed to ultraviolet A (UVA) irradiation inside the machine, and then returned to the patient.

As photopheresis has been used worldwide for more than 30 years, each hospital has developed their own guidelines (e.g. which patients, frequency, etc). Recently, experts in the field have developed a guidance which will now be tested in this study.

ELIGIBILITY:
Inclusion criteria:

* Erythrodermic mycosis fungoides or Sézary Syndrome (T4, N0-3, M0, B0-2) (for staging see table 1)
* World Health Organization (WHO) performance status (PS) 0-2
* Any prior treatment
* With the exception of topical corticosteroids, skin care, itch and pain relieves all prior therapies for MF/SS have to be stopped/completed before registration.
* No specific wash out period prior to registration is defined
* Age ≥ 18, no upper limit
* Measurable disease
* Adequate bone marrow function at time of registration :
* Hemoglobin > 9.0 g/dL (> 5.6 mmol/L);
* White blood cell count > 1 x 109/L (> 1000/mm3) and < 25 x 109/L (< 25,000/mm3);
* Platelet count > 20 x 109/L (> 20,000/mm3);
* Serum creatinine ≤ 1.5 x upper limit of normal (ULN) or estimated glomerular filtration rate (eGFR) according to Modification of Diet in Renal Disease (MDRD) ≥ 50 mL/min
* Serum albumin ≥ 2.8 g/dL.
* Women of child bearing potential (WOCBP) must have a negative serum or urine pregnancy test within 72 hours prior to the initiation of the first study treatment.
* WOCBP should use adequate birth control measures, as defined by the investigator, during the study treatment period and for at least 1 month after the last study treatment. A highly effective method of birth control is defined as those which result in low failure rate (i.e. less than 1% per year) when used consistently and correctly. Such methods include:
* Combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal, transdermal).
* Progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, implantable).
* Intrauterine device (IUD)
* Intrauterine hormone-releasing system (IUS)
* Bilateral tubal occlusion
* Vasectomised partner
* Sexual abstinence (the reliability of sexual abstinence needs to be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient)
* Male patients with pregnant or non-pregnant WOCBP partner should use condom during the study treatment period and for at least 1 month after the last study treatment.
* Female subjects who are breast feeding should discontinue nursing prior to the first dose of study treatment and until 1 month after the last study treatment.
* Before patient registration, written informed consent must be obtained according to international conference on harmonisation/Good clinical practice (ICH/GCP) and national/local regulations.

Exclusion criteria

* History of congestive heart failure (CHF): New York Heart Association (NYHA) Class III (moderate) or Class IV (severe)
* History of any of the following cardiovascular conditions within 6 months prior to registration:
* Unstable angina.
* Clinically significant cardiac arrhythmias.
* Myocardial infarction.
* Poorly controlled hypertension defined at baseline as blood pressure (BP) >150/100 mmHg despite optimal antihypertensive treatment within 7 days of the first dose of study treatment
* Active cancer other than MF/SS. Exceptions:
* Patients with actinic keratoses should not be excluded, treatment should be decided by the treating physician according to local standards of care and be documented in the case report forms (CRFs)
* Patients with non-skin in situ tumors (e.g. mucosal of any site, breast,,…) should be adequately treated prior to study entry.
* Need for any systemic cancer therapy other than ECP at the time of registration according to the treating physician's decision
* History of idiosyncratic or hypersensitivity reaction to methoxsalen, psoralen compounds or any of the excipients
* Aphakia
* History of photosensitive disease like but not limited to porphyria, systemic lupus erythematosus, or albinism.
* Any medical conditions that do not allow extracorporeal volume loss like but not limited to severe cardiac disease, severe anaemia, severe renal disorder
* Previous splenectomy
* Coagulation disorders
* Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-12-01 (Estimated); Primary Completion 2022-09-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Success rate of treatment (photopheresis) | From treatment start up to 9 months for each patient
  The primary endpoint is defined as successful use of photopheresis performed according to the study protocol based on the consensus guidelines.
  At 9 months time point after the initiation of photopheresis, evaluation of each patient will be performed. A patient will be declared a success with respect to the primary endpoint if she/he fulfills:
  1. Patient has received the full protocol treatment
  2. No progressive disease within the first 3 months after of the initiation of photopheresis.
  3. No need for add-on (combination) treatment within the first 3 months after the initiation of photopheresis according to investigators decision.
  4. Not experiencing any medical event (other than progressive disease) necessitating termination of photopheresis or interruption for more than 3 continuous months within the 6 months period

SECONDARY OUTCOMES:
Progression Free Survival, according to EORTC-International Society of Cutaneous Lymphoma (ISCL)-United States Cutaneous Lymphoma Consortium (USCLC) criteria | From the first patient treatment start till 9 months as of LPI
  From treatment start to progression
Best overall response rates, according to EORTC-ISCL-USCLC criteria | From the first patient treatment start till 9 months as of LPI
  Overall response rate is defined as the proportion of patients with global response score equal to complete response (CR) or partial response (PR) according to EORTC-ISCL-USCLC criteria.
  Global Response Score
  CR - Complete disappearance of all clinical evidence of disease; Skin: CR, Nodes/Blood/Viscera: All categories have CR/Not Indicated
  PR - Regression of measurable disease; Skin: CR, Nodes/Blood/Viscera: All categories do not have a CR/ Not Indicated and no category has a PD or Skin: PR, Nodes/Blood/Viscera: No category has a PD and if any category involved at baseline, at least one has a CR or PR
Number of treatment cycles required to obtain remission | From the first patient treatment start till 9 months as of LPI
  Number of treatment cycles (including the add-on therapies) received by patients to obtain remission
Time to response (CR/PR) | From the first patient treatment start till 9 months as of LPI
  From treatment start to progression
Duration of response | From the first patient treatment start till 9 months as of LPI
  From response to progression
Frequency and type of of add-on therapies | From the first patient treatment start till 9 months as of LPI
  Frequency and type of add-on therapies received by patients. The add-on could consist any systemic or skin directed therapies that is considered to be active in or given with the intent to treat MF/SS.
Quality of life measurements | From the first patient treatment start till 9 months as of LPI
  Skin disease-specific Skindex-29 and the Functional Assessment of Cancer Therapy in General (FACT-G)
  SKINDEX-29: Symptoms scale ranging from: Very little, Mild, Moderate, Severe, Extreme
  FACT G: 5-point Likert scale ranging from 0 (Not at all) to 4 (Very much)
Occurrence of adverse events | From the first patient treatment start till 9 months as of LPI
  The study uses the International Common Terminology Criteria for Adverse Events (CTCAE), version 5.0, for adverse event reporting.
Overall survival (OS) | From the first patient treatment start till 3 years as of LPI
  Registration till the date of death from any cause
Time to initiation of add-on therapies | From the first patient treatment start till 9 months as of LPI
  Time to initiation of add-on therapies will be measured from the date of treatment start to the date that add-on therapies initiated

CONTACTS AND LOCATIONS:
Overall Officials: Robert Knobler, Study Chair — Medical University Vienna - General Hospital AKH, Vienna, Austria; Franz Trautinger, Study Chair — Karl Landsteiner University of Health Sciences, University Hospital of St. Poelten, St. Poelten, Austria
Locations (1):
- UniversitaetsSpital Zurich - Division of Dermatology, Zurich, Switzerland